CLINICAL TRIAL: NCT02518438
Title: A Randomized Trial of the Analgesic Efficacy of Wound Infiltration With Tramadol After Cesarean Delivery Under General Anesthesia
Brief Title: The Analgesic Efficacy of Wound Infiltration With Tramadol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, Murat Haliloglu, Medical doctor, Yeditepe University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 190
Record Dates: First submitted 2015-07-08; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Pain
Keywords: Tramadol; Postoperative analgesia; Infiltration; Cesarean section
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- the tramadol group (Active Comparator): A preprepared 20 ml solution (tramadol 2 mgkg-1 within a 0.9% saline solution) was subcutaneously infiltrated after closure of the uterine incision and the rectus fascia.
  Interventions: Drug: Tramadol
- the placebo group (Placebo Comparator): A preprepared 20 ml solution (0,9% saline solution) was subcutaneously infiltrated after closure of the uterine incision and the rectus fascia.

INTERVENTIONS:
Drug: Tramadol — A preprepared 20 ml solution was subcutaneously infiltrated after closure of the uterine incision and the rectus fascia.
  Other Names: Placebo (0,9% saline solution)
  Arms: the tramadol group

SUMMARY:
This double-blind, randomized trial examined whether tramadol wound infiltration decreased postoperative pain following cesarean delivery under general anesthesia or reduced the need for analgesics in the immediate postoperative period. Patients in the tramadol group consumed significantly less morphine at all time intervals than those in the control group. The investigators suggest that the use of wound infiltration with tramadol may be a useful technique in patients who undergo cesarean section under general anesthesia to reduce postoperative pain, improve recovery, and facilitate early contact of mothers with their babies.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparity
* Gestation age between 37-40 weeks
* CS under general anesthesia

Exclusion Criteria:

* Pre-eclampsia
* Cardiovascular problems
* Allergy to any of the study medications
* Chronic preoperative pain
* Regular analgesic use

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure in this study was cumulative morphine consumption. | postoperative 24 hours
  The measure of need for analgesics in the immediate postoperative period in this study was cumulative morphine consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University Hospital, Istanbul, Kozyatagı, Turkey (Türkiye)